CLINICAL TRIAL: NCT06755307
Title: PROBIOTICS FOR TREATING DIAPER DERMATITIS IN CHILDREN - A DOUBLE-BLIND, RANDOMIZED, PLACEBO-CONTROLLED CLINICAL TRIAL
Brief Title: Probiotics for Diaper Dermatitis
Acronym: ProDiaper II
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Maribor (Other)
Responsible Party: Principal Investigator, Sabina Fijan, Assoc. Prof. Dr., University Maribor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UKC-MB-KME-59/22
Record Dates: First submitted 2024-12-23; First posted 2025-01-01 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Diaper Dermatitis
Keywords: diaper dermatitis; probiotics; children
MeSH Terms: conditions — Diaper Rash

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PROBIOTIC (Experimental): Multistrain Probiotic OMNiBiOTiC® Panda containing probiotics and sunflower oil
  Interventions: Dietary Supplement: OMNiBiOTiC® Panda
- Placebo (Placebo Comparator): Placebo containing sunflower oil and maltodextrin
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: OMNiBiOTiC® Panda — Multistrain Probiotic OMNiBiOTiC® Panda containing: Bifidobacterium bifidum W23 Bifidobacterium lactis W51 Bifidobacterium lactis W52 Lactococcus lactis W58 and sunflower oil
  Arms: PROBIOTIC
Other: Placebo — Placebo containing sunflower oil and maltodextrin
  Arms: Placebo

SUMMARY:
The goal of this randomized controlled clinical trial is to determine the effect of the probiotic OMNiBiOTiC® Panda in treating diaper dermatitis in children under the age of two years. The main question it aims to answer is:

Is the probiotic OMNiBiOTiC® Panda effective in reducing the duration of diaper dermatitis in children under the age of two years?

Researchers will compare the probiotic and placebo group to see if the duration of diaper dermatitis is significant among the two groups.

Participants will:

* receive 6 droplets daily of probiotic or placebo for 3 weeks and
* observe and record improvement of diaper rash symptoms each day using a diary.

ELIGIBILITY:
Inclusion Criteria:

* presence of diaper dermatitis
* age less than two years

Exclusion Criteria:

* previous use of probiotics
* age more than two years
* an acute bacterial infection
* chronic disease
* local use of antibiotics in the anogenital region

Ages: 1 Month to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 42 (Estimated)
Dates: Start 2025-08-14 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Duration of diaper dermatis | 3 weeks supplementation
  Comparison of the duration of diaper dermatitis in children younger than two years in both arms via daily the use of the diary.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maribor, Faculty of Health Sciences, Maribor, Slovenia

IPD SHARING:
Plan to Share IPD: No